CLINICAL TRIAL: NCT03549975
Title: Hand Rehabilitation Using Botulinum Toxin and Functional Electrical Stimulation Among Stroke Patients With Limitation of Finger Extension Due to Spasticity- Pilot Study
Brief Title: Hand Rehabilitation Using Botulinum Toxin and Functional Electrical Stimulation-pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager of Department of Neurorehabilitation, National Rehabilitation Center, Seoul, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRC-2016-02-011
Record Dates: First submitted 2018-05-16; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Stroke; Spastic Hemiparesis; Spasticity as Sequela of Stroke
Keywords: stroke; hand; botulinum toxin; functional electrical stimulation
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Botulinum toxin type A injection (Experimental): Botulinum toxin type A injection followed by functional electrical stimulation
  Interventions: Drug: Botulinum Toxin Type A 100 unit/Vial (Product)

INTERVENTIONS:
Drug: Botulinum Toxin Type A 100 unit/Vial (Product) — Botulinum toxin type A injection followed by functional electrical stimulation
  Other Names: functional electrical stimulation

SUMMARY:
The investigator tried to find out possibility of functional improvement using botulinum toxin injection targeting finger flexor spasticity with functional electrical stimulation among chronic stroke patients who did not show any improvement in hand function.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* hemiplegic upper limb spasticity secondary to a unilateral ischemic or hemorrhagic stroke
* fingers and wrist flexor spasticity graded at least 1+ on the Modified Ashworth Scale
* at least 6 months since stroke

Exclusion Criteria:

* fixed contracture
* previous treatment of the upper limb spasticity with neurolytic or surgical procedure
* treatment with botulinum toxin type A in the previous 4 months
* any active device implant
* any neurological disorder, other than stroke causing motor deficits or spasticity
* inability to attend to and/or to cooperate with all outcome measure-related task secondary to cognitive impairment or aphasia
* pregnancy, planned pregnancy, or lactation
* contraindication to botulinum toxin type A

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Change in Box and Block test | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  number of box moved by affected upper extremity
Change of Action Research Arm Test | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  Score of Action Research Arm Test

SECONDARY OUTCOMES:
Muscle strength of finger extensor | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  Medical research council grading of muscle strength
Spasticity of finger extensor | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  Modified ashworth scale of finger flexor
active range of motion of wrist joint | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  active range of motion of wrist joint
Brunnstrom stage of stroke recovery of distal upper extremity | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  Brunnstrom stage of stroke recovery of distal upper extremity. By observing the pattern of participants posture, the stage was scored. The stage ranges from 1 to 6. Higher is better.
Distance from middle finger tip to mid-palmar crease | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  Distance from middle finger tip to mid-palmar crease
Repeated number of finger extension and flexion | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  Repeated number of finger extension and flexion
Quick Disabilities of Arm, Shoulder & Hand | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  Quick Disabilities of Arm, Shoulder & Hand is questionnaire about patients' symptoms as well as ability to perform certain activities in the last week.
  Total score is obtained by summing the each question, and ranges from 0 (no disability) to 100 (most severe disability).
Grading of active thumb opposition | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  Grading of active thumb opposition. It is measured by observing the pattern of thumb opposition.
Grip strength | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  measured by Jamar dynamometer
Active finger extension | baseline, 2 weeks after baseline, 6 weeks after baseline, 10 weeks after baseline
  Active finger extension. It is graded by observation of voluntary finger extension.

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center of Korea